CLINICAL TRIAL: NCT05016089
Title: The Efficacy of a Simplified Pilates Exercise Training in Reducing the Risk of Falling in Hong Kong's Older Adults: A Wait-list Randomised Controlled Trial
Brief Title: Simplified Pilates Training in Older Adults in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18191091
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Aged
Keywords: Efficacy; Simplified Pilates; Wait-list control; Falls prevention; Older adults; Risk of falling; Fall risk factors; Hong Kong

STUDY DESIGN:
Intervention Model Description: A randomised, controlled (wait-list control), and two-armed trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified Pilates exercise group (SPEG) (Experimental): The participants in the SPEG will participate in the 16-style simplified Pilates exercise sessions (about 60 minutes each) in a group (about 10 participants in each group) twice a week for 12 weeks. Each participant will undertake a total of 24 exercise sessions.
  Interventions: Other: The 16-style simplified Pilates exercise programme
- Wait-list control group (WLCG) (Other): The participants in the WLCG will participate in the 16-style simplified Pilates exercise sessions (about 60 minutes each) in a group (about 10 participants in each group) twice a week for 12 weeks after two scheduled assessment sessions and a waiting period of 12 weeks in between. Each participant will undertake a total of 24 exercise sessions.
  Interventions: Other: The 16-style simplified Pilates exercise programme

INTERVENTIONS:
Other: The 16-style simplified Pilates exercise programme — The 16-style simplified Pilates exercise programme was developed by a group of experienced Pilates and rehabilitation experts from our completed pilot work.

SUMMARY:
This study aims to examine the efficacy of the simplified Pilates exercise programme developed by a group of Pilates and rehabilitation experts in Hong Kong to reduce the risk of falling (the physical and psychological risk factors) of Hong Kong's older adults who might be prone to falling. It is hypothesized that a simplified Pilates exercise programme is efficacious in reducing the risk of falling (the physical and psychological risk factors) in Hong Kong's older adults who are at a medium to high risk of falling. There is no updated research that has specifically investigated an expertly designed simplified Pilates exercise programme and no research investigated it in Hong Kong as well. Therefore, this study is novel and important in investigating the efficacy of an expertly designed simplified Pilates exercise programme in Hong Kong's older population specifically developed for reducing the risk of falls. It could increase the intelligent choices of efficacious and easy-to-comply-with fall prevention exercise programmes (the 16-style simplified Pilates exercise programme) for older adults and reduce the impact of falls in the older population. The more the choices of simple and efficacious fall prevention programmes that are available for older adults, the more likely it is that they will be interested in complying with the programme. Consequently, this research could provide evidence of Pilates being used in fall prevention of older adults locally and globally.

DETAILED DESCRIPTION:
This study will be a randomised controlled trial to investigate the efficacy of the simplified Pilates exercise programme (developed by a group of Pilates and rehabilitation experts in Hong Kong in our completed pilot study) by comparing it with the wait-list control.

A total of 60 older adults will be recruited from different collaborating community elderly and rehabilitation centres in Hong Kong using convenience sampling. The inclusion criteria will be the following: (1) age 65 or above and (2) score of less than 24/28 in the Tinetti Performance Oriented Mobility Assessment (POMA). The exclusion criteria will be the following: (1) total score of less than 24 in the Chinese version of the Mini-Mental State Examination (MMSE-C), (2) presence of any untreated cerebral vascular disease, Parkinson's disease, or any other major neurological deficit, (3) presence of any unstable medical condition that can affect safety during the exercise training, and (4) inability to sit and lie down on a Pilates exercise mat on the floor even with assistance.

The participants (N = 60) will be randomly assigned using concealed block randomisation by an independent person through a sealed and opaque envelope system to either the simplified Pilates exercise group (SPEG; n = 30) or the wait-list control group (WLCG; n = 30). A computerised random-number generator will be utilised to prepare an allocation schedule. The participants in the SPEG will partake in exercise sessions (about 60 minutes each) in a group (about 10 participants in each group) twice a week for 12 weeks. Each participant will undertake a total of 24 exercise sessions. All the training sessions will be conducted in Hong Kong by two experienced and certified Pilates trainers under the supervision of a registered physiotherapist. The participants in the SPEG will practise the 16-style simplified Pilates exercise programme. The WLCG will participate in the 16-style simplified Pilates exercise programme after two scheduled assessment sessions and a waiting period of 12 weeks in between.

To examine the efficacy of the exercise programme, the participants of both the SPEG and WLCG will undergo two assessment sessions before training at baseline (T0) and just after the completion of all the exercise sessions (T1). In the baseline assessment (T0), a structural questionnaire will be used to ask the participants for their demographic information, detailed information regarding any previous falls, detailed medical history, use of prescribed drugs, social history, and socio-economic status. Following this, a series of assessments will be conducted to examine their balance ability, which will be measured by the Berg Balance Scale (BBS; primary outcome measure), and other physical and psychological fall risk factors (secondary outcome measures) in the two assessment sessions (T0 & T1). Any adverse events will be reported and tracked. Participants will also be asked to prospectively record the number of falls they have experienced during the time between T0 and T1 using a structural calendar. The frequency of falls (secondary outcome measure) will then be collected at T1.

Balance ability (primary outcome measure) will be assessed using the BBS. Regarding the other physical fall risk factors (secondary outcome measure), flexibility will be measured using the 'sit-and-reach' (S&R) test. A functional gait and balance assessment will be conducted using the POMA and Timed Up and Go (TUG) tests.

On the other hand, for the assessment of the psychological fall risk factors (secondary outcome measure), the MMSE-C will be used as a screening tool to examine the preliminary cognitive function at the beginning of training. Depression levels will be assessed using the Chinese version of the 4-item Geriatric Depression Scale (GDS-4C). Anxiety levels will be measured using the valid and reliable Chinese version of the State-Trait Anxiety Inventory (STAT-SC & STAI-TC). The valid and reliable Chinese version of the Falls Efficacy Scale International [FES-I (Ch)] will be utilised to assess the fear of falling. The valid and reliable Chinese version of the Activities-Specific Balance Confidence Scale [ABC (Ch)] will be used to evaluate balance confidence.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 or above;
2. score of less than 24/28 in the Tinetti Performance Oriented Mobility Assessment (POMA).

Exclusion Criteria:

1. total score of less than 24 in the Chinese version of the Mini-Mental State Examination (MMSE-C);
2. presence of any untreated cerebral vascular disease, Parkinson's disease, or any other major neurological deficit;
3. presence of any unstable medical condition that can affect safety during the exercise training;
4. inability to sit and lie down on a Pilates exercise mat on the floor even with assistance.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Balance Ability | Day 0
  Berg Balance Scale (BBS)
Change from Baseline Balance Ability at 12 weeks | Week 12
  Berg Balance Scale (BBS)

SECONDARY OUTCOMES:
Baseline Flexibility | Day 0
  Sit-and-reach (S&R) test
Change from Baseline Flexibility at 12 weeks | Week 12
  Sit-and-reach (S&R) test
Baseline Functional Gait and Balance Assessment | Day 0
  The Tinetti Performance Oriented Mobility Assessment (POMA)
Change from Baseline Functional Gait and Balance Assessment at 12 weeks | Week 12
  The Tinetti Performance Oriented Mobility Assessment (POMA)
Baseline Functional Gait Assessment | Day 0
  Timed Up and Go (TUG) tests
Change from Baseline Functional Gait Assessment at 12 weeks | Week 12
  Timed Up and Go (TUG) tests
Preliminary Cognitive Function | Day 0
  The Chinese version of the Mini-Mental State Examination (MMSE-C)
Baseline Depression Levels | Day 0
  The Chinese version of the 4-item Geriatric Depression Scale (GDS-4C)
Change from Baseline Depression Levels at 12 weeks | Week 12
  The Chinese version of the 4-item Geriatric Depression Scale (GDS-4C)
Baseline Anxiety Levels | Day 0
  The Chinese version of the State-Trait Anxiety Inventory (STAT-SC & STAI-TC)
Change from Baseline Anxiety Levels at 12 weeks | Week 12
  The Chinese version of the State-Trait Anxiety Inventory (STAT-SC & STAI-TC)
Baseline Fear of Falling | Day 0
  The Chinese version of the Falls Efficacy Scale International [FES-I (Ch)]
Change from Baseline Fear of Falling at 12 weeks | Week 12
  The Chinese version of the Falls Efficacy Scale International [FES-I (Ch)]
Baseline Balance Confidence | Day 0
  The Chinese version of the Activities-Specific Balance Confidence Scale [ABC (Ch)]
Change from Baseline Balance Confidence at 12 weeks | Week 12
  The Chinese version of the Activities-Specific Balance Confidence Scale [ABC (Ch)]
Frequency of falls | Week 12
  Participants will be asked to prospectively record the number of falls they have experienced during the time between Day 0 and Week 12 using a structural calendar. The frequency of falls will be collected at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Thomson Wong, PhD, BScPT, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No